CLINICAL TRIAL: NCT05131217
Title: Effects of Acute Exercise Intensity on Cerebral Blood Flow and Cognitive Function in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jason Allen, Professor of Exercise Physiology at the University of Virginia, Director of the Exercise Physiology Graduate Program & Co-Director of the Applied Metabolism & Physiology Lab, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HSR200454
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Aging Well
Keywords: MCAv; Working Memory; Cognition; Exercise Intensity; Cerebral Blood Flow; HIIT
MeSH Terms: interventions — RE1-silencing transcription factor

STUDY DESIGN:
Intervention Model Description: This is a repeated measures cross-over design, in which all subjects will complete all acute exercise intensity conditions: HIIT, continuous moderate intensity at lactate threshold (LT), and rest (control). The order of the acute treatment bouts will be randomized for each subject over three experimental visits (not counting the screening visit).
Who Masked: Outcomes Assessor
Masking Description: The individual analyzing study data will be blind to subject allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acute bout of Continuous Moderate Intensity Exercise (Experimental)
  Interventions: Other: Acute bout of Continuous Moderate Intensity Exercise
- Acute bout of High Intensity Interval Training (HIIT) (Experimental)
  Interventions: Other: Acute bout of High Intensity Interval Training
- Control (Experimental)
  Interventions: Other: Control

INTERVENTIONS:
Other: Acute bout of Continuous Moderate Intensity Exercise — In this experimental intervention subjects will cycle continuously at moderate intensity (VO2 corresponding to lactate threshold) until a 200 kcal equivalent energy expenditure is reached.
  Arms: Acute bout of Continuous Moderate Intensity Exercise
Other: Acute bout of High Intensity Interval Training — In this experimental invention subjects will alternate between 1 minute of high intensity cycling (watts corresponding to 85% VO2peak) and 1 minute of low intensity cycling (watts corresponding to 35-40% VO2peak) until a 200 kcal equivalent energy expenditure is reached.
  Other Names: HIIT
  Arms: Acute bout of High Intensity Interval Training (HIIT)
Other: Control — In this intervention placebo, subjects will lay down on a flat, soft surface for 30 minutes in a dimly light room. They will not be allowed to use any electronic devices or read during this time to avoid potentially influencing continuous data recording.
  Other Names: Rest
  Arms: Control

SUMMARY:
This study will analyze the influence of acute bout exercise intensities (continuous moderate and HIIT) on middle cerebral artery velocity (MCAv) to identify which intensity elicits the greatest increase in CBF in older adults (65+ yrs). Additionally, this study will help verify positive correlations between MCAv and cognitive function. These findings are important in determining the optimal exercise prescription for increased resilience against the age-related cognitive degradation.

DETAILED DESCRIPTION:
With an increasingly aging population, it is paramount that we further understand the changes that occur during aging, especially those which contribute to cognitive decline. Evidence shows that cognitive function is closely linked to brain blood flow. When comparing cerebral blood flow (CBF) between old and young individuals, older adults appear to have lower baseline levels of CBF. One of the principle determinants of CBF is CO2. Since exercise results in rises in CO2 production, changes in CBF can be monitored. Older adults appear to have diminished changes in CBF compared to younger individuals during moderate intensity exercise. This then leads to the idea that older adults may need a greater exercise stimulus (i.e. HIIT) to see these changes in CBF. However, the effects of HIIT on CBF in older adults is largely unstudied.

Purpose: To analyze the acute influence of HIIT on middle cerebral artery velocity (MCAv) in older adults, and to verify the positive association between MCAv and cognitive function.

Experimental Design: Recruiting 16 healthy adults age 65 and older. The study will require each participant to report to 4 visits: a screening visit, a control, a moderate intensity exercise bout, and a high intensity exercise bout. The order of the experimental visits will be randomized to each subject, and exercise bouts will be work-matched. During the experimental visits, MCAv, end-tidal CO2, MAP, and HR will be measured continuously. Vascular measures such as pulse wave analysis and pulse wave velocity will be taken pre- and post-exercise. Additionally, blood flow through the internal carotid artery and cognitive measures (n-back test) will be measured and administered pre-exercise, and at 15 mins, 30 mins, and 45 mins post-exercise. A two-way repeated measures ANOVA will be used to determine significant differences for time (pre vs. post measures) x condition (control/moderate/HIIT).

Results: In the process of collecting data.

Implications: If the study is successful in its findings, this could change how exercise is prescribed to older adults. It could also lead to the question regarding if a greater exercise stimulus (i.e. SIT) may be even more beneficial for these individuals.

ELIGIBILITY:
Inclusion Criteria:

* 65+ years of age
* Comfortable with experiencing exercise-induced fatigue
* Willingness and ability to comply with scheduled visits and study procedures
* Able to provide consent on their own behalf
* Type 2 Diabetics accepted

Exclusion Criteria:

* Competitive athlete (Recreationally active is okay but no more than 3 days/week of structured exercise)
* VO2max below 18 ml/kg/min in men, 15ml/kg/min in women (minimum thresholds for independent living seniors)
* Inability of study staff to acquire signal from the MCA using TCD
* Diagnosis of mild cognitive impairment, Parkinson's Disease, Alzheimer's Disease, multiple sclerosis, or psychiatric illness (unless mild depression or anxiety)
* History of brain damage/stroke/concussions
* Cardiovascular Disease, Pulmonary Disease, or dependence of supplemental O2
* Type 2 Diabetics who aren't cleared by the study physician during the first screening visit (HbA1C > 8.5%)
* Neuromuscular or musculoskeletal dysfunctions impairing one from cycling
* Changes in vasoactive medication dose or quantity, recently prior to or during the study time course, or inability to maintain regular timed ingestion of vasoactive medication
* Currently involved in Estrogen or Testosterone Replacement Therapy
* Unable to abstain from food consumption (3hrs), caffeine/alcohol consumption (12hrs), and vigorous exercise (24hrs) prior to experimental procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Middle Cerebral Artery Velocity (MCAv) | Measured continuously over the course of each experimental session (i.e. 2-3 hours)
  Blood flow velocity measured in the Middle Cerebral Artery via Transcranial Doppler probe secured to the right temporal window.

SECONDARY OUTCOMES:
Working Memory | 4 individual measurements taken during each experimental session with each session lasting up to about 3 hours. 1 pre-intervention measurement and 3 post-intervention measurements spaced at least 15min apart
  Measured via n-back test (2-back); Subject's will be presented a sequence of letters (25 of them from a base set of 15 letters) one-by-one and will have 3 seconds to indicate whether the letter they see currently matches the letter from 2 frames ago. If there is no match, then they do not need to respond.They will complete three rounds each with a different sequence. Accuracy score (%) = correct inputs/# of stimuli, averaged across 3 blocks.
Internal Carotid Artery (ICA) Diameter | 4 individual measurements taken during each experimental session with each session lasting up to about 3 hours. 1 pre-intervention measurement and 3 post-intervention measurements spaced at least 15min apart
  Measured via Ultrasound; diameter will be measured as the peak of the pulse wave
Internal Carotid Artery (ICA) Pulse Velocity | 4 individual measurements taken during each experimental session with each session lasting up to about 3 hours. 1 pre-intervention measurement and 3 post-intervention measurements spaced at least 15min apart
  Measured via Ultrasound; velocity will be assessed at the peak of each pulse wave

OTHER OUTCOMES:
Heart Rate | Measured continuously over the course of each experimental session (i.e. 2-3 hours)
  Measured via three-lead ECG
End Tidal CO2 (ETCO2) | Measured continuously over the course of each experimental session (i.e. 2-3 hours)
  Measured via Capnograph; connected nasal cannulas are placed in the nostrils and respiration will be assessed continuously
Mean Arterial Pressure (MAP) | Measured continuously over the course of each experimental session (i.e. 2-3 hours)
  Measured via Finger photoplethysmography (Non-Invasive Blood Pressure; NIBP), pressure cuffs on the subjects fingers will take continual blood pressure readings via continual inflation and deflation
Augmentation Index (AI) | 4 individual measurements taken during each experimental session with each session lasting up to about 3 hours. 1 pre-intervention measurement and 3 post-intervention measurements spaced at least 15min apart
  Measured via Pulse Wave Analysis; a SphygmoCor device probe will be held on carotid artery and pulse wave will be analyzed
Pulse Wave Velocity (Brachial-Femoral) | 4 individual measurements taken during each experimental session with each session lasting up to about 3 hours. 1 pre-intervention measurement and 3 post-intervention measurements spaced at least 15min apart
  Measured via SphygmoCor; distances between brachial artery and femoral artery will be taken for calibration, cuffs at the brachial and femoral arteries will inflate and SphygmoCor will take pulse wave measurements
Internal Carotid Artery (ICA) Distensibility | 4 individual measurements taken during each experimental session with each session lasting up to about 3 hours. 1 pre-intervention measurement and 3 post-intervention measurements spaced at least 15min apart
  Measured via Ultrasound; diameter will be measured during both systole and diastole

CONTACTS AND LOCATIONS:
Overall Officials: Jason Allen, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia; Kinesiology Labs, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thudium M, Heinze I, Ellerkmann RK, Hilbert T. Cerebral Function and Perfusion during Cardiopulmonary Bypass: A Plea for a Multimodal Monitoring Approach. Heart Surg Forum. 2018 Jan 31;21(1):E028-E035. doi: 10.1532/hsf.1894. PMID 29485961
- [Background] Shoemaker LN, Wilson LC, Lucas SJE, Machado L, Thomas KN, Cotter JD. Swimming-related effects on cerebrovascular and cognitive function. Physiol Rep. 2019 Oct;7(20):e14247. doi: 10.14814/phy2.14247. PMID 31637867
- [Background] Alexandrov AV, Sloan MA, Wong LK, Douville C, Razumovsky AY, Koroshetz WJ, Kaps M, Tegeler CH; American Society of Neuroimaging Practice Guidelines Committee. Practice standards for transcranial Doppler ultrasound: part I--test performance. J Neuroimaging. 2007 Jan;17(1):11-8. doi: 10.1111/j.1552-6569.2006.00088.x. PMID 17238867
- [Background] Burley CV, Francis ST, Whittaker AC, Mullinger KJ, Lucas SJE. Measuring resting cerebral haemodynamics using MRI arterial spin labelling and transcranial Doppler ultrasound: Comparison in younger and older adults. Brain Behav. 2021 Jul;11(7):e02126. doi: 10.1002/brb3.2126. Epub 2021 May 25. PMID 34032379
- [Background] Fan JL, Nogueira RC, Brassard P, Rickards CA, Page M, Nasr N, Tzeng YC. Integrative physiological assessment of cerebral hemodynamics and metabolism in acute ischemic stroke. J Cereb Blood Flow Metab. 2022 Mar;42(3):454-470. doi: 10.1177/0271678X211033732. Epub 2021 Jul 26. PMID 34304623
- [Background] Klein T, Sanders M, Wollseiffen P, Carnahan H, Abeln V, Askew CD, Claassen JA, Schneider S. Transient cerebral blood flow responses during microgravity. Life Sci Space Res (Amst). 2020 May;25:66-71. doi: 10.1016/j.lssr.2020.03.003. Epub 2020 Mar 19. PMID 32414494
- [Background] Loe H, Rognmo O, Saltin B, Wisloff U. Aerobic capacity reference data in 3816 healthy men and women 20-90 years. PLoS One. 2013 May 15;8(5):e64319. doi: 10.1371/journal.pone.0064319. Print 2013. PMID 23691196
- [Background] Ogoh S, Ainslie PN. Cerebral blood flow during exercise: mechanisms of regulation. J Appl Physiol (1985). 2009 Nov;107(5):1370-80. doi: 10.1152/japplphysiol.00573.2009. Epub 2009 Sep 3. PMID 19729591
- [Background] Settakis G, Lengyel A, Molnar C, Bereczki D, Csiba L, Fulesdi B. Transcranial Doppler study of the cerebral hemodynamic changes during breath-holding and hyperventilation tests. J Neuroimaging. 2002 Jul;12(3):252-8. PMID 12116744
- [Background] Shephard RJ. Maximal oxygen intake and independence in old age. Br J Sports Med. 2009 May;43(5):342-6. doi: 10.1136/bjsm.2007.044800. Epub 2008 Apr 10. PMID 18403414
- [Background] Jones-Muhammad M, Warrington JP. Redefining the cerebral autoregulatory range of blood pressures: Not as wide as previously reported. Physiol Rep. 2021 Sep;9(17):e15006. doi: 10.14814/phy2.15006. PMID 34435458
- [Background] Keating CJ, Parraga Montilla JA, Latorre Roman PA, Moreno Del Castillo R. Comparison of High-Intensity Interval Training to Moderate-Intensity Continuous Training in Older Adults: A Systematic Review. J Aging Phys Act. 2020 Apr 16;28(5):798-807. doi: 10.1123/japa.2019-0111. Print 2020 Oct 1. PMID 32303000
- [Result] Smith KJ, Ainslie PN. Regulation of cerebral blood flow and metabolism during exercise. Exp Physiol. 2017 Nov 1;102(11):1356-1371. doi: 10.1113/EP086249. Epub 2017 Sep 30. PMID 28786150
- [Result] Calverley TA, Ogoh S, Marley CJ, Steggall M, Marchi N, Brassard P, Lucas SJE, Cotter JD, Roig M, Ainslie PN, Wisloff U, Bailey DM. HIITing the brain with exercise: mechanisms, consequences and practical recommendations. J Physiol. 2020 Jul;598(13):2513-2530. doi: 10.1113/JP275021. Epub 2020 Jun 1. PMID 32347544
- [Result] Ogoh S, Tsukamoto H, Hirasawa A, Hasegawa H, Hirose N, Hashimoto T. The effect of changes in cerebral blood flow on cognitive function during exercise. Physiol Rep. 2014 Sep 28;2(9):e12163. doi: 10.14814/phy2.12163. Print 2014 Sep 1. PMID 25263210
- [Result] Siasos G, Athanasiou D, Terzis G, Stasinaki A, Oikonomou E, Tsitkanou S, Dimitropoulos S, Kolokytha T, Tzirogiannis K, Giannaki A, Tousoulis D. The Acute Impact of Different Types of Aerobic Exercise on Arterial Wave Reflections and Inflammation. Cardiology. 2016;135(2):81-6. doi: 10.1159/000445993. Epub 2016 Jun 10. PMID 27287855
- [Result] Ward JL, Craig JC, Liu Y, Vidoni ED, Maletsky R, Poole DC, Billinger SA. Effect of healthy aging and sex on middle cerebral artery blood velocity dynamics during moderate-intensity exercise. Am J Physiol Heart Circ Physiol. 2018 Sep 1;315(3):H492-H501. doi: 10.1152/ajpheart.00129.2018. Epub 2018 May 18. PMID 29775407
- [Result] Labrecque L, Drapeau A, Rahimaly K, Imhoff S, Billaut F, Brassard P. Comparable blood velocity changes in middle and posterior cerebral arteries during and following acute high-intensity exercise in young fit women. Physiol Rep. 2020 May;8(9):e14430. doi: 10.14814/phy2.14430. PMID 32342622
- [Result] Barnes JN, Taylor JL, Kluck BN, Johnson CP, Joyner MJ. Cerebrovascular reactivity is associated with maximal aerobic capacity in healthy older adults. J Appl Physiol (1985). 2013 May 15;114(10):1383-7. doi: 10.1152/japplphysiol.01258.2012. Epub 2013 Mar 7. PMID 23471946
- [Result] Billinger SA, Craig JC, Kwapiszeski SJ, Sisante JV, Vidoni ED, Maletsky R, Poole DC. Dynamics of middle cerebral artery blood flow velocity during moderate-intensity exercise. J Appl Physiol (1985). 2017 May 1;122(5):1125-1133. doi: 10.1152/japplphysiol.00995.2016. Epub 2017 Mar 9. PMID 28280106
- [Result] Coverdale NS, Lalande S, Perrotta A, Shoemaker JK. Heterogeneous patterns of vasoreactivity in the middle cerebral and internal carotid arteries. Am J Physiol Heart Circ Physiol. 2015 May 1;308(9):H1030-8. doi: 10.1152/ajpheart.00761.2014. Epub 2015 Feb 27. PMID 25724496
- [Result] Gonzalez-Alonso J, Dalsgaard MK, Osada T, Volianitis S, Dawson EA, Yoshiga CC, Secher NH. Brain and central haemodynamics and oxygenation during maximal exercise in humans. J Physiol. 2004 May 15;557(Pt 1):331-42. doi: 10.1113/jphysiol.2004.060574. Epub 2004 Mar 5. PMID 15004212
- [Result] Hoiland RL, Smith KJ, Carter HH, Lewis NCS, Tymko MM, Wildfong KW, Bain AR, Green DJ, Ainslie PN. Shear-mediated dilation of the internal carotid artery occurs independent of hypercapnia. Am J Physiol Heart Circ Physiol. 2017 Jul 1;313(1):H24-H31. doi: 10.1152/ajpheart.00119.2017. Epub 2017 Apr 7. PMID 28389602
- [Result] Lefferts WK, DeBlois JP, Barreira TV, Heffernan KS. Neurovascular coupling during cognitive activity in adults with controlled hypertension. J Appl Physiol (1985). 2018 Dec 1;125(6):1906-1916. doi: 10.1152/japplphysiol.00100.2018. Epub 2018 Jul 26. PMID 30048202
- [Result] Lefferts WK, DeBlois JP, Receno CN, Barreira TV, Brutsaert TD, Carhart RL, Heffernan KS. Effects of acute aerobic exercise on arterial stiffness and cerebrovascular pulsatility in adults with and without hypertension. J Hypertens. 2018 Aug;36(8):1743-1752. doi: 10.1097/HJH.0000000000001752. PMID 29677054
- [Result] Lie SL, Hisdal J, Hoiseth LO. Cerebral blood flow velocity during simultaneous changes in mean arterial pressure and cardiac output in healthy volunteers. Eur J Appl Physiol. 2021 Aug;121(8):2207-2217. doi: 10.1007/s00421-021-04693-6. Epub 2021 Apr 22. PMID 33890157
- [Result] Lucas SJ, Ainslie PN, Murrell CJ, Thomas KN, Franz EA, Cotter JD. Effect of age on exercise-induced alterations in cognitive executive function: relationship to cerebral perfusion. Exp Gerontol. 2012 Aug;47(8):541-51. doi: 10.1016/j.exger.2011.12.002. Epub 2012 Jan 2. PMID 22230488
- [Result] Moraine JJ, Lamotte M, Berre J, Niset G, Leduc A, Naeije R. Relationship of middle cerebral artery blood flow velocity to intensity during dynamic exercise in normal subjects. Eur J Appl Physiol Occup Physiol. 1993;67(1):35-8. doi: 10.1007/BF00377701. PMID 8375362
- [Result] Ogoh S. Relationship between cognitive function and regulation of cerebral blood flow. J Physiol Sci. 2017 May;67(3):345-351. doi: 10.1007/s12576-017-0525-0. Epub 2017 Feb 3. PMID 28155036
- [Result] Olivo G, Nilsson J, Garzon B, Lebedev A, Wahlin A, Tarassova O, Ekblom M, Lovden M. Immediate effects of a single session of physical exercise on cognition and cerebral blood flow: A randomized controlled study of older adults. Neuroimage. 2021 Jan 15;225:117500. doi: 10.1016/j.neuroimage.2020.117500. Epub 2020 Oct 24. PMID 33169699
- [Result] Weaver SR, Skinner BD, Furlong R, Lucas RAI, Cable NT, Rendeiro C, McGettrick HM, Lucas SJE. Cerebral Hemodynamic and Neurotrophic Factor Responses Are Dependent on the Type of Exercise. Front Physiol. 2021 Jan 21;11:609935. doi: 10.3389/fphys.2020.609935. eCollection 2020. PMID 33551835
- [Result] Belfort MA, Saade GR, Snabes M, Dunn R, Moise KJ Jr, Cruz A, Young R. Hormonal status affects the reactivity of the cerebral vasculature. Am J Obstet Gynecol. 1995 Apr;172(4 Pt 1):1273-8. doi: 10.1016/0002-9378(95)91492-7. PMID 7726269
- [Result] Jones RD, Hugh Jones T, Channer KS. The influence of testosterone upon vascular reactivity. Eur J Endocrinol. 2004 Jul;151(1):29-37. doi: 10.1530/eje.0.1510029. PMID 15248819
- [Result] Fulesdi B, Limburg M, Bereczki D, Kaplar M, Molnar C, Kappelmayer J, Neuwirth G, Csiba L. Cerebrovascular reactivity and reserve capacity in type II diabetes mellitus. J Diabetes Complications. 1999 Jul-Aug;13(4):191-9. doi: 10.1016/s1056-8727(99)00044-6. PMID 10616858
- [Result] Coetsee C, Terblanche E. The effect of three different exercise training modalities on cognitive and physical function in a healthy older population. Eur Rev Aging Phys Act. 2017 Aug 10;14:13. doi: 10.1186/s11556-017-0183-5. eCollection 2017. PMID 28811842